CLINICAL TRIAL: NCT06830044
Title: A Randomized, Double-Blind, Placebo-controlled Multicenter Study to Assess the Efficacy and Safety of Milsaperidone as Adjunctive Therapy in the Treatment of Patients With Major Depressive Disorder
Brief Title: Evaluation of Efficacy and Safety of Milsaperidone as Adjunctive Therapy in Patients With Major Depressive Disorder
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-VHX-896-3201
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-02

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Milsaperidone (Experimental)
  Interventions: Drug: Milsaperidone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Milsaperidone — Oral milsaperidone
  Other Names: VHX-896
  Arms: Milsaperidone
Drug: Placebo — Oral placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and safety of milsaperidone compared to placebo as adjunctive therapy in patients with Major Depressive Disorder

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient 18 to 65 years of age, inclusive;
* Meets DSM-5-TR criteria for MDD
* Currently having an inadequate response to antidepressant therapy as confirmed by the Investigator using the Antidepressant Treatment Response Questionnaire (ATRQ)

Exclusion Criteria:

* Within the patients lifetime, has a confirmed DSM-5-TR psychiatric diagnosis other than MDD
* Within 6 months of Screening, has a confirmed DSM-5-TR psychiatric diagnosis other than MDD
* Within 12 months of Screening, has had any other psychiatric condition (other than MDD) that has been the main focus of treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) | 6 weeks
  The MADRS is a clinician-rated 10 item scale. Individual item scores are summed for a total possible score of 0 to 60 with a higher score indicating increased severity of depressive symptoms.

CONTACTS AND LOCATIONS:
Locations (19):
- United States (15):
  - Vanda Investigational Site, Little Rock, Arkansas
  - Vanda Investigational Site, Garden Grove, California
  - Vanda Investigational Site, Orange, California
  - Vanda Investigational Site, San Jose, California
  - Vanda Investigational Site, Colorado Springs, Colorado
  - Vanda Investigational Site, Fort Myers, Florida
  - Vanda Investigational Site, Miami, Florida
  - Vanda Investigational Site, Tampa, Florida
  - Vanda Investigational Site, Chicago, Illinois
  - Vanda Investigational Site, Saint Charles, Missouri
  - Vanda Investigational Site, Las Vegas, Nevada
  - Vanda Investigational Site, Staten Island, New York
  - Vanda Investigational Site, Media, Pennsylvania
  - Vanda Investigational Site, Richardson, Texas
  - Vanda Investigational Site, Witchita Falls, Texas
- Bulgaria (2):
  - Vanda Investigational Site, Sofia
  - Vanda Investigational Site, Varna
- Czechia (2):
  - Vanda Investigational Site, Brno
  - Vanda Investigational Site, Prague

IPD SHARING:
Plan to Share IPD: No